CLINICAL TRIAL: NCT06900023
Title: The BEACON Trial: Diagnostic Tools for Breast Lymphedema After Treatment for Breast Cancer
Acronym: BEACON
Status: Enrolling by invitation | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Cheryl Brunelle, Physical Therapy Clinical Specialist, Associate Director, MGH Lymphedema Research Program, Massachusetts General Hospital
Other Study IDs: 23412
Record Dates: First submitted 2025-02-25; First posted 2025-03-28 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Breast Edema; Breast Lymphedema; Lymphedema, Breast Cancer; Lymphedema
Keywords: Breast Edema; Breast Swelling; Breast Lymphedema; Breast Edema Screening; Breast swelling after breast cancer
MeSH Terms: conditions — Breast Cancer Lymphedema; Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants with breast edema: N=15: This group will contain women who report breast edema and have been diagnosed with breast edema through clinical examination
- Participants without breast edema: N=15: These participants do not report a history of breast edema and do not have a history of breast edema.

SUMMARY:
The goal of this observational study is to learn if participants agree to take part in the study, if the methods we are using for the study are feasible for the participants and the researchers, and to study how well two tools (tissue dielectric constant and ultrasound) measure breast edema after breast conserving surgery for breast cancer.

Participants who agree to be in the study will be asked to come in for one appointment of approximately two hours. All data will be collected during this one visit. Participants will be asked to fill out two questionnaires regarding their symptoms, and one questionnaire regarding their surgical scar. The research staff will conduct a clinical examination, measure breast edema using ultrasound and tissue dielectric constant, measure arm volume with the perometer and fluid with the SOZO, and take photographs of both breasts.

DETAILED DESCRIPTION:
The goal of this observational study is to learn if the study protocol is feasible, if we can accrue participants easily, and to determine how well two tools (tissue dielectric constant and ultrasound) identify breast edema after breast conserving surgery for breast cancer.

Participants will be asked to attend one appointment in which all data will be collected. This will include questionnaires regarding symptoms, clinical examination, measurement of breast edema using two tools (ultrasound and tissue dielectric constant), measurement with the perometer and SOZO, and clinical photographs.

ELIGIBILITY:
All participants must meet the following inclusion criteria:

* Be a female between the ages of 18 and 85 years.
* Have undergone breast conserving surgery +/- LN removal (sentinel lymph node biopsy (SLNB) or axillary lymph node dissection (ALND)
* Have no residual cancer in the breast after definitive breast surgery
* Have been treated with radiation therapy and have completed breast cancer treatment (excluding Herceptin and hormonal treatments) at MGH greater than or equal to 3 months ago.
* Be able to read and understand English
* Understand the proposed study and be willing and fully able to comply with the study procedures
* Be a willing participant and be capable of giving and has given informed written consent for entry into the study

EXCLUSION CRITERIA

Participants will be excluded if they:

* Have bilateral BC
* Have metastatic or inflammatory BC
* Will be excluded from the SOZO measurement of the study if they have implanted cardiac devices or neurostimulators
* Have any medical condition that may result in breast swelling;

  * Uncontrolled congestive cardiac failure,
  * Arteriovenous haemodialysis,
  * Current infection or cellulitis of either breast.
* Be pregnant or currently breast feeding.
* Have a known over-active thyroid or known benign thyroid tumour

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women screened for lymphedema in the MGH Lymphedema Research Program Prospective Screening Program; and/or women treated in physical or occupational therapy for breast cancer-related conditions after breast conserving surgery.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Tissue Dielectric Constant | Baseline
  A TDC interbreast ratio ≥ 1.28 in any quadrant will be used as an indicator of breast lymphedema
Breast Ultrasound | Baseline
  Skin thickness >1.60 mm in superior and lateral quadrants, >2.0 mm in the medial and inferior quadrants will be used as an indicator of breast lymphedema.

SECONDARY OUTCOMES:
Patient-Reported Outcome Measures | Baseline
  Breast Cancer Treatment Outcome Scale (BCTOS-12) Minimum Score = 12, Maximum Score = 48 Higher score indicates worse outcome
Patient-Reported Outcome Measures | Baseline
  Breast-Q Version 2.0 Breast Conserving Therapy Module, Postoperative Scales i. Psychosocial Well-Being (min score 10, max score 50), higher score indicating better outcome
Scar Assessment Tool | Baseline
  Patient and Observer Scar Scale Linear Scar Version 3.0
Clinical Examination of Lymphedema of the Upper Extremity Clinical Exam Tool | Baseline
  This is a validated measure used to administer clinical examination of the breast, trunk and upper extremity for lymphedema
Clinical Examination - Pitting Edema | Baseline
  The following will be assessed:
  * Each breast quadrant: Presence or absence of pitting edema
  * The participant is placed in supine. The examiner's thumb is placed firmly on the participant's skin, applying sustained pressure to the skin and superficial tissue for one minute. Upon release of the pressure, an indentation of the tissue at the test site is defined as pitting and is recorded as Yes in the relevant quadrant. If there is no change in the tissue, record No to pitting oedema.
Clinical Examination - Peau d'orange | Baseline
  The following will be assessed:
  * Each breast quadrant, lateral chest wall and inframammary tissues: Presence or absence of peau d'orange
  * The participant is positioned sitting. The examiner slightly compresses the breast tissue between their first finger and thumb to look for the orange peel appearance to the skin. A light can be shone tangentially across the breast to assist in identifying peau d'orange.
Clinical Examination - Tissue fibrosis | Baseline
  The following will be assessed:
  * Each breast quadrant: Presence or absence of tissue fibrosis
  * The participant is placed in supine. The examiner uses their first finger and thumb to palpate the tissue and gently pinch the tissue to assess for any tissue thickening, increased firmness or density and/or tissue retraction or fixation, compared to the equivalent tissue on the unaffected side. If the participant has had surgery on the unaffected breast (e.g. breast reduction), the tissue in the quadrant most distal to the incision site is used as the comparator tissue. N/A is marked in the table for the unaffected breast, unless the participant has had surgery on the unaffected side and tissue fibrosis is detected as a result compared to other quadrants of the unaffected breast.
Clinical Examination - Tenderness to palpation | Baseline
  The following will be assessed:
  * Each breast quadrant: Presence or absence of tenderness to palpation.
  * The examiner will lightly palpate the tissue of each breast quadrant to see if the participant reports any pain or tenderness. Deep palpation, particularly medially in the breast, may cause tenderness in the costochondral cartilages.
Clinical Examination - Erythema | Baseline
  The following will be assessed:
  - Each breast quadrant: Presence or absence of erythema (redness of the skin)
Clinical Examination - Scar localization | Baseline
  The following will be assessed:
  - Scar measurements for the breast and axillary scars, including location (quadrant, distance from the center of the nipple to the center of the scar), scar length, width and orientation (vertical, horizontal, oblique or radial).
Clinical Examination - Visual fullness | Baseline
  The following will be assessed:
  - Lateral chest wall and inframammary tissue: The examiner will record presence or absence of visual fullness
Clinical Examination - Stemmer sign | Baseline
  The following will be assessed:
  - Lateral chest wall and inframammary tissue: Presence or absence of the Stemmer sign. The Stemmer sign is a physical examination finding used to diagnose lymphedema. If the examiner cannot pinch the skin then this positive finding is associated with lymphedema. The Stemmer sign has been found to be a sensitive predictor for primary and secondary lymphedema with moderate specificity (Goss JA, Greene AK. Sensitivity and Specificity of the Stemmer Sign for Lymphedema: A Clinical Lymphoscintigraphic Study. Plast Reconstr Surg Glob Open. 2019 Jun 25;7(6):e2295. doi: 10.1097/GOX.0000000000002295. PMID: 31624689; PMCID: PMC6635205)
Clinical Examination - Tissue thickening | Baseline
  The following will be assessed by the examiner:
  - Nipple and nipple-areolar complex: Tissue thickening on the side of surgery as compared to the unaffected side
Clinical Examination - Skin color changes | Baseline
  The following will be assessed by the examiner:
  - Nipple and nipple-areolar complex: Skin color changes as compared to the unaffected side (lighter, darker, same)
Patient-Reported Outcome Measures | Baseline
  Breast-Q Version 2.0 Breast Conserving Therapy Module, Postoperative Scales ii. Sexual Well-Being (min score 6, max score 30), higher score indicating better outcome
Patient-Reported Outcome Measures | Baseline
  Breast-Q Version 2.0 Breast Conserving Therapy Module, Postoperative Scales iii. Satisfaction with Breasts (min score 11, max score 44), higher score indicating better outcome
Patient-Reported Outcome Measures | Baseline
  Breast-Q Version 2.0 Breast Conserving Therapy Module, Postoperative Scales iv. Physical Well-Being: Chest (min score 10, max score 30), higher score indicating better outcome
Patient-Reported Outcome Measures | Baseline
  Breast-Q Version 2.0 Breast Conserving Therapy Module, Postoperative Scales v. Adverse Effects of Radiation (min score 6, max score 18), higher score indicating better outcome
Patient-Reported Outcome Measures | Baseline
  Breast-Q Version 2.0 Breast Conserving Therapy Module, Postoperative Scales vi. Satisfaction with Information - Breast Surgeon (min score 12, max score 48), higher score indicating better outcome

OTHER OUTCOMES:
Perometry | Baseline
  Perometry will be undertaken per clinical protocol to screen for arm lymphedema
Bioimpedance Spectroscopy (SOZO) | Baseline
  Bioimpedance Spectroscopy will be undertaken per clinical protocol
Clinical Photographs | Baseline
  Clinical photographs of each breast, repeated for the right and then the left breast, taken per study protocol 5 positions each side, including a close up photo of the breast and surgical scar.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Brunelle, MScPT, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No